CLINICAL TRIAL: NCT00967538
Title: Safety and Efficacy of Etanercept in Patients With Moderate to Severe Plaque Psoriasis Who Have Shown an Unsatisfactory Response to Adalimumab or Infliximab
Brief Title: Safety and Efficacy of Etanercept in Patients With Psoriasis Who Failed to Respond to Other Biologic Treatments
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Innovaderm Research Inc. (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Inno-6011; CA-2009-0004
Record Dates: First submitted 2009-08-26; First posted 2009-08-28 (Estimated); Last update posted 2014-07-24 (Estimated); Status verified 2014-07

CONDITIONS: Psoriasis
Keywords: psoriasis; etanercept; efficacy; response; anti-TNF alpha; treatment efficacy
MeSH Terms: conditions — Psoriasis | interventions — Etanercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Etanercept (Experimental): All patients will receive etanercept 50 mg twice a week for 12 weeks followed by 50 mg once a week for an additional 12 weeks.
  Interventions: Drug: etanercept 50 mg

INTERVENTIONS:
Drug: etanercept 50 mg — All patients will receive etanercept 50 mg twice a week for 12 weeks followed by 50 mg once a week for an additional 12 weeks.
  Other Names: Enbrel

SUMMARY:
The purpose of this study is to evaluate safety and efficacy of etanercept in patients with psoriasis who had an unsatisfactory response to adalimumab and infliximab.

ELIGIBILITY:
Inclusion Criteria:

* Patient has plaque psoriasis and has shown an unsatisfactory response to adalimumab. Unsatisfactory response is defined as patients who failed to reach a PGA of clear or almost clear (PGA of 0 or 1) following at least 12 weeks with adalimumab at 40 mg EOW; OR
* Patient has plaque psoriasis and has lost his/her satisfactory response to adalimumab. Loss of satisfactory response is defined as patients treated with adalimumab 40 mg EOW for at least 12 weeks, who achieved a PGA of clear or almost clear (PGA of 0 or 1) but lost this PGA response (increase in PGA to 2, 3, 4 or 5) at any time after 12 weeks of adalimumab; OR
* Patient has plaque psoriasis and has lost his/her satisfactory response to infliximab. Loss of satisfactory response is defined as patients treated with at least 3 infliximab infusions at 5 mg/kg, who achieved a PGA of clear or almost clear (PGA of 0 or 1) but lost this PGA response (increase in PGA to 2, 3, 4 or 5) at any time after the 3rd infusion of infliximab;
* Patient's age is 18 to 80 years old;
* Patient has PGA of 3 or more at Day 0;
* Patient has BSA of 3% or more at Day 0;
* Patient has psoriasis severe enough to be eligible to systemic therapy;
* Unless surgically sterile (or at least 1 year post-menopausal for women), or abstinent, patient (male or female) is willing to use an effective method of contraception for at least 30 days before Day 0 and until at least 1 month after the last drug administration;
* Patient capable of giving informed consent;
* Patient with normal or non clinically significant chest X-ray within 6 months prior to Day 0;
* Patient with negative Purified Protein Derivative (PPD) or Quantiferon TB Gold test within 90 days prior to Day 0;
* Female patients of childbearing potential have a negative serum pregnancy test;
* Patient is able to start etanercept per the approved product monograph.

Exclusion Criteria:

* Patient has used topical steroids, topical tar preparations, or other anti-psoriatic preparations within the two weeks prior to Day 0 or during the study period, unless patient used topical therapy during the last 4 weeks of the period when the patient lost their satisfactory response to adalimumab or infliximab or when the patient failed to achieve a satisfactory response to adalimumab;
* Patient has presence of erythrodermic, pustular or guttate psoriasis;
* Patient has had significant infections within the 30 days prior to Day 0;
* Patient has received investigational drugs within the four weeks prior to screening or during the study period;
* Patient has been treated with systemic anti-psoriatic drugs such as steroids, retinoids, cyclosporine, PUVA therapy or methotrexate within the four weeks prior to Day 0 or during the study period;
* Patient received systemic antibiotics within the four weeks prior to Day 0;
* Patient has been treated with ultraviolet light therapy (UVB, nbUVB) within the two weeks prior to Day 0 or during the study period;
* Patient has used adalimumab or infliximab within 14 days of Day 0 or during the study period;
* Patient has used other biologic agents for the treatment of psoriasis besides etanercept 8 weeks prior to Day 0 or during the study period;
* Patient has had an allergic reaction to adalimumab, infliximab or etanercept;
* Patient has an unstable or serious medical condition as defined by the investigator or presence of any significant medical condition that might cause this study to be detrimental to the patient;
* Uncontrolled or severe comorbidities such as poorly controlled diabetes mellitus, NYHA class III or IV heart failure, history of myocardial infarction or cerebrovascular accident or transient ischemic attack within three months of screening visit; unstable angina pectoris; uncontrolled hypertension, oxygen-dependent severe pulmonary disease;
* Patient has a known sero-positivity for HIV virus or history of any other immunosuppressive disease;
* Patient has active or chronic Hepatitis B or C;
* Patient has any mycobacterial disease, patient with a chest X-Ray suggestive of tuberculosis or patient taking anti-tuberculosis medication;
* Patient has a known hypersensitivity to etanercept or one of its components;
* Patient has received a live attenuated vaccine within the 12 weeks prior to Day 0 or plans to receive one during the study;
* Current pregnancy or lactation;
* At the investigator

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2009-09; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who reach a Physician's Global Assessment (PGA) of clear or almost clear after 12 and 24 weeks of etanercept for patients who have shown an unsatisfactory response to adalimumab 40 mg every other week (EOW). | 24 weeks

SECONDARY OUTCOMES:
Proportion of patients who reach a PGA of clear or almost clear after 12 and 24 weeks of etanercept for patients who have lost their satisfactory response to adalimumab 40 mg EOW. | 24 weeks
Proportion of patients who reach a PGA of clear or almost clear after 12 and 24 weeks of etanercept for patients who have lost their satisfactory response to infliximab. | 24 weeks
Mean Body Surface Area (BSA) after 12 weeks and 24 weeks of etanercept for patients who have lost their satisfactory response to infliximab. | 24 weeks
Mean BSA after 12 weeks and 24 weeks of etanercept for patients who have lost their satisfactory response to adalimumab 40 mg EOW. | 24 weeks
Mean BSA after 12 and 24 weeks of etanercept for patients who have shown an unsatisfactory response to adalimumab 40 mg EOW. | 24 weeks
Mean Psoriasis Area and Severity Index (PASI) score after 12 weeks and 24 weeks of etanercept for patients who have lost their satisfactory response to infliximab. | 24 weeks
Mean PASI score after 12 weeks and 24 weeks of etanercept for patients who have lost their satisfactory response to adalimumab 40 mg EOW. | 24 weeks
Mean PASI score after 12 and 24 weeks of etanercept for patients who have shown an unsatisfactory response to adalimumab 40 mg EOW. | 24 weeks
Safety of etanercept in patients who have shown an unsatisfactory response to adalimumab, who have lost their satisfactory response to adalimumab or who have lost their satisfactory response to infliximab. | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ronald B Vender, MD, Principal Investigator — Dermatrials Research; Robert Bissonnette, MD, Principal Investigator — Innovaderm Research Inc.
Locations (16):
- Canada (16):
  - Kirk Barber Research, Calgary, Alberta
  - PerCuro Clinical Research Ltd, Victoria, British Columbia
  - Winnipeg Clinic Dermatology Research, Winnipeg, Manitoba
  - Nexus Clinical Research, St. John's, Newfoundland and Labrador
  - New Lab Clinical Research, St. John's, Newfoundland and Labrador
  - Eastern Canada Cutaneous Research Associates Ltd, Halifax, Nova Scotia
  - Sudbury Skin Clinic, Greater Sudbury, Ontario
  - Dermatrials Research, Hamilton, Ontario
  - Mediprobe Research Inc., London, Ontario
  - Lynderm research Inc., Markham, Ontario
  - Dermatology Associates, North York, Ontario
  - Dr. Jay Brian Taradash, Toronto, Ontario
  - Innovaderm Research Inc., Montreal, Quebec
  - Siena Medical Research, Montreal, Quebec
  - Centre de Recherches Dermatologiques du Quebec Metropolitain, Québec, Quebec
  - Clinique Esthetique Dr Isabelle Delorme, Saint-Hyacinthe, Quebec